CLINICAL TRIAL: NCT03029559
Title: Intermittent Hypoxia and Inspiratory Threshold Loading as Strategies to Enhance Inspiratory Muscle Function
Brief Title: Intermittent Hypoxia and Inspiratory Threshold Loading to Enhance Inspiratory Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201601878
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Intermittent Hypoxia
Keywords: Inspiratory threshold loading

STUDY DESIGN:
Intervention Model Description: Latin square, repeated measures design to study the effects of IH administered alone and in combination with inspiratory threshold loading on the above stated respiratory parameters.
Who Masked: Participant
Masking Description: We will use a Latin square, repeated measures design which will consist of 12 subjects participating in the following four experimental conditions: There will be an interval of 1 week between each of the four conditions, which will serve as a washout period.
  1. IH+ITL: Subjects will be exposed to a session of IH (45 minutes, 2 minutes of hypoxia alternating with 1 minute of hyperoxia) followed by 5 sets of ITL at 80%MIP (10 breaths per set).
  2. IH: Subjects will only be exposed to a session of intermittent hypoxia.
  3. Sham IH +ITL: Subjects will be exposed to a single 45-minute session of sham IH (normoxia). This will consist of the subject breathing room air (FiO2=21%) through a 4 way valve connected to the hypoxicator. Exposure to normoxia will be followed by 5 sets of ITL at 80%MIP (10 breaths per set).
  4. Sham IH: Subjects will be exposed to a single 45-minute session of sham IH (normoxia) alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IH + ITL (Experimental): Subjects will be exposed to a session of Intermittent hypoxia (IH) (45 minutes, 2 minutes of hypoxia alternating with 1 minute of hyperoxia) followed by 5 sets of Inspiratory threshold loading (ITL) at 80%MIP (10 breaths per set).
  Interventions: Other: Intermittent Hypoxia; Other: Inspiratory Threshold Loading
- Intermittent hypoxia (IH) (Experimental): Subjects will only be exposed to a session of intermittent hypoxia.
  Interventions: Other: Intermittent Hypoxia
- Sham IH + ITL (Experimental): Sham Intermittent Hypoxia + Inspiratory threshold loading (ITL) subjects will be exposed to a single 45-minute session of sham IH (normoxia). This will consist of the subject breathing room air (FiO2=21%) through a 4 way valve connected to the hypoxicator. Exposure to normoxia will be followed by 5 sets of ITL at 80%MIP (10 breaths per set).
  Interventions: Other: Inspiratory Threshold Loading; Other: Sham Intermittent Hypoxia
- Sham IH (Sham Comparator): Sham intermittent hypoxia subjects will be exposed to a single 45-minute session of sham IH alone.
  Interventions: Other: Sham Intermittent Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — A single session of IH will last for 45 minutes and will consist of alternating phases of hypoxia(FiO2 :9%-11%) and hyperoxia (FiO2 :22%-38%).
  Each hypoxic interval will last for 2 minutes whereas the hyperoxic interval lasts for 1 minute each (15, two-minute episodes of hypoxia and 15, one-minute episodes of hyperoxia).
  Other Names: IH
  Arms: IH + ITL; Intermittent hypoxia (IH)
Other: Inspiratory Threshold Loading — Subjects will undergo inspiratory threshold loading using a commercially available Threshold IMT device (Power breathe®). ITL will be administered at an intensity of 80% of the individual's maximal inspiratory pressure (MIP). The subjects will be instructed to take 10 deep, forceful breaths through the threshold device followed by at least 2 minutes of rest. The process will be repeated 4 more times for a total of 5 sets of 10 breaths each.
  Other Names: ITL
  Arms: IH + ITL; Sham IH + ITL
Other: Sham Intermittent Hypoxia — Subjects will be exposed to a session of sham Intermittent hypoxia.This will consist of breathing room air for 45 minutes through a hypoxicator.
  Other Names: Normoxia
  Arms: Sham IH; Sham IH + ITL

SUMMARY:
Rehabilitation approaches introduce a stimulus to a motor system, with the goal to enhance motor function to patients. For example, exposure to brief and intermittent episodes of mild hypoxia has shown to strengthen synaptic pathways to respiratory and skeletal muscle motor neurons. In humans with spinal cord injury, exposure to intermittent hypoxia (IH) alone or in combination with rehabilitative strategies has shown enhanced motor function. Another strategy known as inspiratory threshold loading, which involves breathing against pressure threshold loads, results in improved inspiratory muscle strength. Although there is evidence supporting the use of IH alone or in combination with other rehabilitative strategies in improving motor function in humans, the impact of exposure to IH or IH with inspiratory threshold loading on inspiratory muscle function and ventilation in humans is unknown.

DETAILED DESCRIPTION:
Investigators will test whether exposure to IH alone and in combination with inspiratory threshold loading (ITL) will result in increased inspiratory muscle strength and ventilation.

Investigators will use a Latin square, repeated measures design which will consist of 12 subjects participating in four experimental conditions.There will be an interval of 1 week between each of the four conditions, which will serve as a washout period.

At the end of each of the 5 sessions, the subjects will rest in a reclining chair for 15 minutes while their heart rate, blood pressure, oxygen saturation and breathing are monitored. Subjects that have a blood systolic blood pressure > 140 or diastolic pressure > 90 or SPO2 < 92% will be asked to remain in the laboratory for 15 additional minutes and the vital signs will be repeated. If the blood pressure and/or peripheral capillary oxygen saturation (SPO2) remain outside of the criteria mentioned above, the subject will be instructed to seek assessment by their health provider and the incident will be reported to the Institutional Review Board. Subjects will also be asked to report any discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Participating in three or fewer musculoskeletal strength training sessions per week at an intensity equivalent to 7-10 on the Modified Borg's scale
* Participating in three or fewer cardiovascular endurance training sessions per week at an intensity equivalent to 7-10 on the Modified Borg's scale

Exclusion Criteria:

* Diagnosis of cardiovascular disease (Hypertension, arrhythmias, coronary artery disease, congenital and valvar heart diseases)
* Diagnosis of neuromuscular disease
* Diagnosis of any neurological disease
* Presence of concurrent medical illness including infection, fractures
* Diagnosis of obstructive sleep apnea
* Diagnosis of obstructive/restrictive lung disease
* Diagnosis of exercise induced asthma
* Forced expiratory volume at one second/forced vital capacity (FVC) <80% and/or FVC<80% of predicted value indicating airway obstruction
* Subjects on prednisolone therapy or selective serotonin reuptake inhibitor (SSRI) therapy will be excluded from the study.
* Diagnosis of epilepsy or history of seizures and attention deficit disorders
* Pregnancy
* Diabetes
* History of coagulation disorders
* History of chronic pain
* Body mass index(BMI)> 35kg/m2
* Subjects on prescription medicines such as beta blockers and other drugs that are prescribed in any of the exclusionary disorders listed above.
* Any other factor that in the investigators' opinions would prevent response to training or create an unsafe condition for the subject.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure will be measured across all groups | Change between 15, 30, and 60 minutes
  Maximal Inspiratory Pressure(MIP) which is a measure of inspiratory muscle strength will be measured as the MIP recorded at the mouth by a pressure manometer. Subjects will be seated upright in a comfortable chair and the nose occluded with clips. After exhaling to residual volume (RV), subjects place their lips around the mouthpiece and inspire as forcefully as possible for at least three seconds. Repeated measurements will be taken, with a 1- to 2-min rest between trials, until three measurements are obtained within 5% variability. Of these three values, the best MIP will be recorded.
Ventilatory responses to inspiratory loading will be measured across all groups | Change between 15, 30, and 60 minutes
  Subjects will be asked to breathe as forcefully as possible against a inspiratory load( 2-4 sets of 5 repetitions) of either 40% of their maximal inspiratory pressure(MIP) or at 41CmH2O (lowest of the two as the maximum resistance offered by the device is 41CmH2O) using a inspiratory muscle training (IMT) device. During this task, a respiratory monitor will be connected to the IMT device. Parameters such as the inspiratory flow, volume and pressure generated by the subjects while breathing against the load will be recorded. Imposed work of breathing (WOBi) will be calculated as a product of the pressure generated and the inspired tidal volume when breathing against a fixed load (40%MIP).
Mouth occlusion pressure (P0.1) will be measured across all groups | Change between 15, 30, and 60 minutes
  To record P0.1, the subjects will breathe through a mouth piece connected to a 2 way respiratory valve in a closed circuit. As the subjects breathe through the circuit, the inspiratory valve will be manually occluded during the expiratory phase and the occlusion will be maintained till the end of next inspiration. Occlusion will be random in order to prevent the subjects from getting conscious about the occlusions. The circuit is connected to the respiratory monitor and the negative pressure recorded in the first 100 milliseconds of the occluded breath will be recorded as the subject's P0.1.
  3 such recordings will be obtained and the highest pressure amongst the 3 trials will be considered for analysis.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) will be measured across all groups | Change between 15, 30, and 60 minutes
  Heart Rate Variability (HRV): HRV will be assessed to determine the autonomic response to intermittent hypoxia. HRV will be measured using a 3 lead ECG and HRV recording kit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Martin, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States